CLINICAL TRIAL: NCT01520974
Title: ProBiora3 Oral Care Probiotics Usage
Brief Title: Effect of an Oral Probiotic Tablet on Oral Bacteria and Clinical Measurements (ProBiora3)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oragenics, Inc. (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ORA.2011.PB3
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Oral Health

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic tablet (Active Comparator)
  Interventions: Other: ProBiora3 mints
- Placebo tablet (Placebo Comparator): Comparison tablet without the probiotic bacteria
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Other: ProBiora3 mints — Probiotic mint tablet taken once daily for 12 weeks containing ProBiora3, a combination of three known healthy bacteria
  Other Names: EvoraPlus; EvoraPro
  Arms: Probiotic tablet
Other: Placebo tablet — Mint tablet taken once daily for 12 weeks without the ProBiora3 combination of three known healthy bacteria
  Other Names: placebo
  Arms: Placebo tablet

SUMMARY:
The purpose of this study is to determine if an oral probiotic tablet taken once a day for twelve weeks can decrease the numbers of bacteria that are associated with tooth decay and gum disease in a dentally healthy, young adult population.

DETAILED DESCRIPTION:
There are over 500 types of bacteria in the mouth. Most of these bacteria do not cause disease. However, some mouth bacteria can cause tooth decay and gum disease. The purpose of a probiotic tablet for the mouth is to put known healthy bacteria in the mouth. This study will compare the effect of the probiotic tablet on the levels of harmful or disease causing bacteria in the mouth to a placebo tablet that does not contain any probiotic bacteria.

ELIGIBILITY:
Inclusion Criteria:

* minimum of 20 teeth, with only a few fillings
* good general health
* willing to use an appropriate method of birth control during the study
* measurable levels of Streptococcus mutans and one or more of the selected periodontal pathogens

Exclusion Criteria:

* chronic or acute illness such as heart disease, diabetes, cancer, hepatitis (liver disease) or HIV positive
* radiation therapy or systemic cancer treatment (chemotherapy)
* require antibiotics for dental treatment
* pregnant or planning to become pregnant during the study period

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Enumeration of S. mutans in saliva and seven periodontal pathogens in subgingival plaque | 12 weeks
  Quantitative RT-PCR analyses for S. mutans in saliva, and A. actinomycetemcomitans, P. intermedia, T. forsythia, F. nucleatum, C. rectus, and E. corrodens in subgingival dental plaque.

SECONDARY OUTCOMES:
Breath odor | 12 weeks
  Halimeter used to evaluate breath odor
Teeth whiteness | 12 weeks
  Teeth whiteness measured with VITA Toothguide 3D-MASTER

CONTACTS AND LOCATIONS:
Overall Officials: Whasun O Chung, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Scool of Dentistry, Regional Clinical Dental Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Zahradnik RT, Magnusson I, Walker C, McDonell E, Hillman CH, Hillman JD. Preliminary assessment of safety and effectiveness in humans of ProBiora3, a probiotic mouthwash. J Appl Microbiol. 2009 Aug;107(2):682-90. doi: 10.1111/j.1365-2672.2009.04243.x. Epub 2009 Mar 30. PMID 19486429